CLINICAL TRIAL: NCT04198506
Title: Viral Load Guided Immunosuppression After Lung Transplantation, an Open-label, Randomized, Controlled, Parallel-group, Multicenter Trial
Brief Title: Viral Load Guided Immunosuppression After Lung Transplantation
Acronym: VIGILung
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KKS-256; 2019-001770-29 (EudraCT Number)
Record Dates: First submitted 2019-12-05; First posted 2019-12-13 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Transplantation Lung
Keywords: lung transplantation; dosing immunosuppression; toxicity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tailored tacrolimus dosing (Experimental): Tacrolimus doses will be adapted according to tacrolimus blood level (conventional therapeutic drug monitoring - TDM) and additionally depending on TTV viral load.
  Interventions: Other: Tailored tacrolimus dosing
- Conventional tacrolimus dosing (Active Comparator): Tacrolimus doses will be adapted according to tacrolimus blood level (conventional therapeutic drug monitoring - TDM).
  Interventions: Other: Conventional tacrolimus dosing

INTERVENTIONS:
Other: Tailored tacrolimus dosing — Tacrolimus doses will be adapted according to tacrolimus blood level (conventional therapeutic drug monitoring -TDM) and additionally depending on TTV viral load.
  Arms: Tailored tacrolimus dosing
Other: Conventional tacrolimus dosing — Tacrolimus doses will be adapted according to tacrolimus blood level (conventional therapeutic drug monitoring - TDM).
  Arms: Conventional tacrolimus dosing

SUMMARY:
The VIGILung study is an open-label, randomized, multicenter trial in lung transplant recipients to investigate the safety and efficacy of personalized immunosuppression guided by DNA monitoring of Torque-Teno-Virus (TTV). The aim of the study is to investigate an individual adaptation of the calcineurin inhibitor tacrolimus (tailored calcineurin inhibitor dosing) by a non-invasive biomarker (TTV viral load in whole blood) compared to conventional calcineurin inhibitor dosing. Indicator for toxicity will be the glomerular filtration rate (GFR), which will be estimated using the CKD-EPI formula. 250 patients (age ≥ 18 years) with 21 to 42 days after de novo lung transplantation (bilateral or combined) will be screened as possible subjects eligible for the study. N = 144 patients have to be randomized in two study arms. In Arm 1 tacrolimus doses will be adapted according to the tacrolimus blood level (conventional therapeutic drug monitoring - TDM) and additionally depending on TTV viral load. In Arm 2 tacrolimus doses will be adapted according to TDM.

ELIGIBILITY:
Inclusion Criteria:

1. patients 21 to 42 days after primary de novo lung transplantation (bilateral including combined)
2. age ≥ 18 years
3. tacrolimus based immunosuppression
4. written informed consent
5. detectable TTV load at randomization (>2,7 log 10)
6. negative serum pregnancy test in women of childbearing potential.
7. women of childbearing capacity must agree to maintain highly effective methods of contraception by practicing abstinence or by using at least two methods of birth control from the date of consent through the end of the study. If abstinence is not practiced, a combination of hormonal contraceptive (oral, injectable or implants) and a barrier method (condom, diaphragm with a vaginal spermicidal agent) has to be used.

Exclusion Criteria:

1. patients after unilateral or re-do lung transplantation
2. history or high-risk of obstructive airway complications after lung transplantation
3. respiratory failure (need for oxygen therapy or ventilation at screening after lung transplantation)
4. inability to undergo transbronchial biopsy
5. advanced kidney failure (GFR CKD-EPI <30 ml/min/1.73m2 at inclusion and/or current renal replacement therapy at inclusion or randomization
6. advanced liver cirrhosis (CHILD-Pugh Score C) after lung transplantation
7. fluctuating tacrolimus drug levels (less than 20% in target range after transplantation)
8. symptoms of significant mental illness and with inability to cooperate or communicate with the investigator.
9. unlikeliness to comply with the study requirements
10. HIV positivity
11. evidence of unsolved drug or alcohol addiction
12. breastfeeding women
13. simultaneous participation in other clinical trials if not permitted by the steering committee

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2020-08-05 (Actual); Primary Completion 2025-03-07 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
ΔGFR change of the glomerular filtration rate GFR | Between randomization and 12 months thereafter
  The primary efficacy endpoint ΔGFR is defined as the change of the glomerular filtration rate GFR between randomization and 12 months thereafter. GFR will be estimated using the CKD-EPI formula.

SECONDARY OUTCOMES:
GFR (CKD-EPI) | 1 and 2 months after transplantation (screening visits) and 0, 3, 6, 9 and 12 months after randomization
  Glomerular filtration rate (the Chronic Kidney Disease Epidemiology Collaboration - CKD-EPI) formula
GFR (Cystatin) | At randomization and 12 months after randomization
  Glomerular filtration rate (Cystatin)
proportion of patients with biopsy-proven acute cellular rejection (grade A1 or higher) | Between randomization and 12 months after randomization
  Proportion of patients with biopsy-proven acute cellular rejection (grade A1 or higher), between randomization and 12 months after randomization
proportion of patients with an episode of biopsy-proven lymphocytic bronchitis (grade B1R or higher) | Between randomization and 12 months after randomization
  proportion of patients with an episode of biopsy-proven lymphocytic bronchitis (grade B1R or higher)
proportion of patients with cytomegalovirus (CMV)-infection and number of CMV-disease episodes | Between randomization and 12 months after randomization
  proportion of patients with cytomegalovirus (CMV)-infection and number of CMV-disease
proportion of patients with community-acquired respiratory viral infection (CARV) | Between randomization and 12 months after randomization
  proportion of patients with community-acquired respiratory viral infection (CARV)
proportion of patients with fungal and bacterial infections | Between randomization and 12 months after randomization
  proportion of patients with fungal and bacterial infections
proportion of patients with any of the above mentioned infections | Between randomization and 12 months after randomization
  proportion of patients with any of the above mentioned infections
proportion of patients with unscheduled or emergency hospitalizations | Between randomization and 12 months after randomization
  proportion of patients with unscheduled or emergency hospitalizations
proportion of patients with ICU admissions | Between randomization and 12 months after randomization
  proportion of patients with ICU admissions
quality of life (EQ-5D visual analog scale) | 1 and 2 months after transplantation (screening visits) and 0, 3, 6, 9 and 12 months after randomization
  European Quality of Life 5 Dimensions - EQ-5D
proportion of patients with new or progressive malignancy | Between randomization and 12 months after randomization
  proportion of patients with new or progressive malignancy
tacrolimus trough levels | 1 and 2 months after transplantation (screening visits) and 0, 3, 6, 9 and 12 months after randomization
  tacrolimus trough levels
daily tacrolimus dose [mg] | 1 and 2 months after transplantation (screening visits) and 0, 3, 6, 9 and 12 months after randomization
  daily tacrolimus dose [mg]
proportion of patients with increased/unchanged/decreased (compared to previous visit) target trough levels of tacrolimus | 1 and 2 months after transplantation (screening visits) and 0, 3, 6, 9 and 12 months after randomization
  proportion of patients with increased/unchanged/decreased (compared to previous visit)
exercise capacity measured by the percent predicted distance achieved in the 6-minute walk test (6-MWT) | at randomization and 12 months thereafter
  exercise capacity measured by the percent predicted distance achieved in the 6-minute walk test (6-MWT)
CD4-Lymphocytes counts | 0, 6 and 12 months after randomization
  CD4-Lymphocytes counts
proportion of patients with presence of donor specific antibodies | 0, 6 and 12 months after randomization
  proportion of patients with presence of donor specific antibodies
FEV1 in % baseline value | 1 and 2 months after transplantation (screening visits) and 0, 3, 6, 9 and 12 months after randomization
  FEV1 in % baseline value
incidence of chronic lung allograft dysfunction | Between randomization and 12 months thereafter
  incidence of chronic lung allograft dysfunction
IgG-level | 0, 6 and 12 months after randomization
  IgG-level
proportion of patients with rescue immunotherapy (defined by the use of ATG, Rituximab, Alemtuzumab, plasma exchange, immunoadsorption) | Between randomization and 12 months thereafter
  proportion of patients with rescue immunotherapy (defined by the use of ATG, Rituximab, Alemtuzumab, plasma exchange, immunoadsorption)
time from randomization to graft loss (defined as re-do transplantation or death) | randomization until 12 months thereafter
  time from randomization to graft loss (defined as re-do transplantation or death)

CONTACTS AND LOCATIONS:
Overall Officials: Jens Gottlieb, Prof. MD, Principal Investigator — Klinik für Pneumologie OE 6870, Medizinische Hochschule Hannover (MHH)
Locations (2):
- Medizinische Universität Wien, Klinische Abteilung für Thoraxchirurgie, Vienna, Austria
- Klinik für Pneumologie OE 6870, Medizinische Hochschule Hannover, Hanover, Germany

IPD SHARING:
Plan to Share IPD: Yes
All proposals of scientific question dealing with the data of the VIGLung-trial have to be approved and released by the steering committee of the trial.
Time Frame: data will be available Begin: one year after publication of results. End: maximum ten years after publication of results
Access Criteria: Approval and release by the steering committee

REFERENCES:
- [Result] Gottlieb J, Reuss A, Mayer K, Weide K, Schade-Brittinger C, Hoyer S, Jaksch P. Viral load-guided immunosuppression after lung transplantation (VIGILung)-study protocol for a randomized controlled trial. Trials. 2021 Jan 11;22(1):48. doi: 10.1186/s13063-020-04985-w. PMID 33430927